CLINICAL TRIAL: NCT01753986
Title: Impact of Brief Substance Use Intervention on Substance Use and Intimate Partner Violence
Brief Title: Alcohol Use and Relationships - III
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1210-005
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Intimate Partner Violence; Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Ethanol; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Alcohol Intervention plus Standard Batterer intervention (Experimental): Brief Alcohol Intervention plus 40 hours of Standard Batterer intervention
  Interventions: Behavioral: Brief Alcohol Intervention plus Standard Batterer Intervention
- General Health Improvement plus Standard batterer intervention (Placebo Comparator): General Health Improvement Intervention plus 40 hours of Standard Batterer intervention
  Interventions: Behavioral: General Health Improvement Intervention plus Standard Batterer Intervention

INTERVENTIONS:
Behavioral: Brief Alcohol Intervention plus Standard Batterer Intervention — Brief Alcohol Intervention plus 40 hours or Standard Batterer Intervention
  Arms: Brief Alcohol Intervention plus Standard Batterer intervention
Behavioral: General Health Improvement Intervention plus Standard Batterer Intervention — General Health Improvement Intervention plus 40 hours of Standard Batterer Intervention
  Arms: General Health Improvement plus Standard batterer intervention

SUMMARY:
The investigators hypothesize that individuals receiving the brief substance use intervention will have better substance use and intimate partner violence outcomes than individuals receiving the general health improvement intervention. All participants receive standard batterer intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participation in Batterer Intervention Program in RI
* Hazardous Drinking

Exclusion Criteria:

* drinks too much

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
lower levels of intimate partner violence | one year
  lower levels of any violence and severe intimate partner violence (psychological, physical, sexual, injuries)

SECONDARY OUTCOMES:
lower levels of substance use (alcohol and drug) | one year

OTHER OUTCOMES:
fewer arrests for violence recidivism | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States